CLINICAL TRIAL: NCT00162500
Title: A Novel Vaccine for the Treatment of MUC1-expressing Tumor Malignancies
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Vaxil Therapeutics Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 191203-HMO-CTIL
Record Dates: First submitted 2005-09-11; First posted 2005-09-13 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2005-09

CONDITIONS: Multiple Myeloma; Tumors
Keywords: Metastatic solid tumors
MeSH Terms: conditions — Multiple Myeloma; Neoplasms | interventions — Protein Subunit Vaccines

INTERVENTIONS:
Biological: Peptide Vaccine (MUC-1)

SUMMARY:
Rationale:

ImMucin was shown to be able to induce a robust cellular immune response mediated via both CD4+ and CD8+ T lymphocytes and therefore, could potentially be more effective in the majority of the target population.

Purpose:

The purpose of this study is to evaluate the safety and initial efficacy of ImMucin, a novel peptide vaccine in metastatic tumors expressing the MUC-1 Tumor Associated Antigen (TAA).

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a histological or cytological diagnosis of metastatic disease expressing the MUC-1. Patients must have metastatic disease and have failed at least one regimen of standard based chemotherapy for metastatic disease such as:

  * Renal Cell Carcinoma (RCC),
  * Transitional Cell Carcinoma (TCC),
  * Prostate,
  * Breast,
  * Ovary,
  * Non-small cell lung,
  * Colon,
  * Multiple myeloma and
  * Pancreatic.
* Patients must be >18 years of age, consenting to participation in the study.
* Patients must have at least one site of measurable tumor or measurable tumor marker.

Exclusion Criteria:

* Patients receiving any immunosuppressive treatment that could negate development of an effective immune response to the vaccine.
* Subjects with prior irradiation to a field that includes more than 25% of their lymph nodes and bone marrow likely to be immunosuppressed will be excluded. However, patients who had standard pelvic field radiation such as adjuvant therapy for rectal cancer are not excluded.
* Pregnant and breast feeding women will be excluded. Premenopausal women who are not practicing or willing to practice adequate birth control methods for a period of 3 months after treatment will be excluded.
* Patients with brain metastases.
* Patients with active infection.
* Patients with HIV hepatitis B surface antigen (HBS Ag) and hepatitis C virus (HCV) positive patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)

PRIMARY OUTCOMES:
Determine the safety and tolerability of vaccination comprising the ImMucin vaccine
combined with Granulocyte Macrophage-Colony Stimulating Factor (GM-CSF), in patients
with multiple myeloma and other MUC-1 antigen-expressing metastatic carcinomas

SECONDARY OUTCOMES:
Determine objective anti-tumor response in patients treated with this regimen;
Determine immune response in patients treated with this regimen

CONTACTS AND LOCATIONS:
Overall Officials: Shimon Slavin, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel